CLINICAL TRIAL: NCT06218745
Title: Prediction Model for Postoperative Acute Kidney Injury in Patients Undergoing Lung Transplantation Using Machine Learning: a Retrospective Cohort Study
Brief Title: Prediction Model for Postoperative AKI in Patients Undergoing Lung Transplantation Using Machine Learning
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Assistant professor for fund, Pusan National University Yangsan Hospital
Other Study IDs: 55-2024-003
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplantation
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: General anesthesia — General anesthesia using 2% propofol, and remifentanil for lung transplantation

SUMMARY:
Since 1963, lung transplantation progress has surged due to immunosuppressive agent advancements. In 2004, 1,815 global lung transplantations were reported. Elderly recipients face impaired lung function and health instability, leading to potential respiratory complications post-surgery.

Postoperative acute renal injury (AKI) can cause temporary or chronic dysfunction, increasing hospitalization, complications, and additional treatment needs. Various factors contribute to postoperative renal dysfunction after lung transplantation, including sustained hypoperfusion, bleeding, heart failure, acute myocardial infarction, pulmonary embolism, sepsis, and medications. Retrospective analysis of adult lung transplant patients' records aims to explore characteristics, anesthesia methods, intraoperative tests, and postoperative acute renal dysfunction, analyzing incidence and risk factors to develop a machine learning predictive model.

DETAILED DESCRIPTION:
Since the first report of lung transplantation in humans in 1963, there has been rapid progress in both the quantity and quality of lung transplantation, driven by the significant advancements in immunosuppressive agents since the mid-1990s. In 2004, a total of 1,815 lung transplantations were reported worldwide. Patients undergoing lung transplantation are often elderly and face not only impaired lung function but also overall health instability, leading to the potential occurrence of respiratory complications post-surgery, even with successful lung transplantation outcomes.

Postoperative acute renal injury (AKI) can result in temporary or even chronic renal dysfunction. AKI following surgery can lead to an increase in hospitalization duration, complications, and the need for additional treatment. Various factors are associated with postoperative renal dysfunction after lung transplantation, including sustained hypoperfusion, hypoperfusion related to intraoperative and postoperative bleeding, heart failure, acute myocardial infarction, pulmonary embolism, sepsis, and more. Medications related to renal dysfunction include those associated with thrombosis or embolism, such as aminoglycosides, amphotericin B, non-steroidal anti-inflammatory drugs (NSAIDs), proton-pump inhibitors, contrast agents, and others. Additionally, graft-versus-host disease is known to be related to renal dysfunction.

The retrospective analysis of medical records from adult patients who underwent lung transplantation aims to investigate patient characteristics, anesthesia methods, intraoperative tests, and the occurrence of postoperative acute renal dysfunction. The goal is to analyze the incidence and risk factors of postoperative renal dysfunction and develop a predictive model through machine learning.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older who underwent lung transplantation for end-stage lung disease

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 years of age or older who underwent lung transplantation for end-stage lung disease
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury (AKI) | Within 48 hours after lung transplantation
  Diagnosis of postoperative AKI is based on the change in serum creatinine concentration within 48 hours after surgery.
  Stage 1: An increase in serum creatinine of ≥ 0.3 mg/dL from baseline or a 1.5-2 times increase (≥ 1.5-2 times).
  Stage 2: An increase in serum creatinine of > 2-3 times from baseline (> 2-3 times).
  Stage 3: An increase in serum creatinine of ≥ 3 times from baseline or an increase to ≥ 4.0 mg/dL from baseline (≥ 4.0 mg/dL, only applicable if it increases by at least 0.5 mg/dL acutely), or initiation of renal replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, Principal Investigator — Department of Anesthesia and Pain Medicine, School of Medicine, Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No